CLINICAL TRIAL: NCT03315182
Title: Phase I/II Gene Transfer Clinical Trial of rAAV9.CMV.hNAGLU for Mucopolysaccharidosis (MPS) IIIB
Brief Title: Gene Transfer Clinical Trial for Mucopolysaccharidosis (MPS) IIIB
Acronym: MPSIIIB
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Abeona has decided to discontinue development activities for Product ABO-101 due to a lack of drug supply and for business reasons unrelated to the product safety profile and/or signs of efficacy
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-002
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Mucopolysaccharidosis Type 3 B
Keywords: MPS IIIB; Sanfilippo Syndrome B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Intervention Model Description: This is a dose escalation trial that will begin with the minimal efficacious dose as determined by preclinical studies and approved by the FDA. During the course of the trial, if safety is shown the dose will be escalated according to the clinical protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Low Dose) rAAV9.CMV.hNAGLU (Experimental): Subjects will receive a single infusion:
  • Cohort 1 (Low Dose): 2 X 10E13 vg/kg (n=2 participants)
  Interventions: Biological: rAAV9.CMV.hNAGLU
- Cohort 2 (Med Dose) rAAV9.CMV.hNAGLU (Experimental): Subjects will receive a single infusion:
  • Cohort 2 (Med Dose): 5 X 10E13 vg/kg (n=4-5 participants)
  Interventions: Biological: rAAV9.CMV.hNAGLU
- Cohort 3 (High Dose) rAAV9.CMV.hNAGLU (Experimental): Subjects will receive a single infusion:
  • Cohort 3 (High Dose): 1 X 10E14 vg/kg (n=4-8 participants)
  Interventions: Biological: rAAV9.CMV.hNAGLU

INTERVENTIONS:
Biological: rAAV9.CMV.hNAGLU — Adeno-associated virus serotype 9 carrying the human NAGLU gene under the control of a CMV enhancer/promoter (rAAV9.CMV.hNAGLU) will be delivered one-time through a venous catheter inserted into a peripheral limb vein.

SUMMARY:
Open-label, dose-escalation clinical trial of rAAV9.CMV.hNAGLU injected intravenously through a peripheral limb vein

DETAILED DESCRIPTION:
Adeno-associated virus serotype 9 carrying the human NAGLU gene under the control of a CMV enhancer/promoter (rAAV9.CMV.hNAGLU) will be delivered one-time through a venous catheter inserted into a peripheral limb vein. A tapering course of prophylactic enteral prednisone or prednisolone will be administered for a period of at least two months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPSIIIB by both of the following two methods:

  * No detectable or significantly reduced NAGLU enzyme activity by plasma.
  * Genomic DNA analysis demonstrating homozygous or compound heterozygous mutations in the NAGLU gene
* Age: From Birth to 2 years or children older than 2 years with a minimum cognitive Development Quotient (DQ) of 60 or above (calculated by Bayley Scales of Infant and Toddler Development - Third Edition)

Exclusion Criteria:

* Inability to participate in the clinical evaluation as determined by Principal Investigator
* Identification of two nonsense or null variants on genetic testing of the NAGLU gene
* Has evidence of an attenuated phenotype of MPS IIIB
* Presence of a concomitant medical condition that precludes lumbar puncture or use of anesthetics
* Active viral infection based on clinical observations as infections by Adenoviruses, Epstein-Barr Virus, Cytomegalovirus, Respiratory Syncytial Virus
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer , or precludes the child from participating in the protocol assessments and follow up as autoimmune diseases requiring immunosuppression, such as juvenile rheumatoid arthritis or idiopathic thrombocytopenia purpura
* Subjects with total anti-AAV9 antibody titers ≥ 1:100 as determined by ELISA binding immunoassay
* Subjects with a positive response for the ELISPOT for T-cell responses to AAV9
* Serology consistent with exposure to HIV, or serology consistent with active hepatitis B or C infection
* Bleeding disorder or any other medical condition or circumstance in which a lumbar puncture (for collection of CSF) is contraindicated according to local institutional policy
* Visual or hearing impairment sufficient to preclude cooperation with neurodevelopmental testing
* Uncontrolled seizure disorder
* Any item (braces, etc.) which would exclude the subject from being able to undergo MRI according to local institutional policy
* Any other situation that precludes the subject from undergoing procedures required in this study
* Subjects with cardiomyopathy or significant congenital heart abnormalities
* The presence of significant non-MPS IlIB related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
* Abnormal laboratory values Grade 2 or higher as defined in CTCAE v4.0 for GGT, total bilirubin, creatinine, hemoglobin, WBC count, platelet count, PT and aPTT
* Female participant who is pregnant or demonstrates a positive urine or serum result at screening assessment (if applicable).
* Any vaccination with viral attenuated vaccines less than 30 days prior to the scheduled date of treatment (and use of prednisolone)
* Previous treatment by Haematopoietic Stem Cell transplantation
* Previous participation in a gene/cell therapy or ERT clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Age Equivalent Developmental score (calculated by the Mullen Scales of Early Learning or the Kaufman Assessment Battery for Children Second Edition, based on developmental age) compared with Natural History Study data | 24 months
Product safety as defined by the incidence, type and severity of treatment-related adverse events and serious adverse events | 24 Months

SECONDARY OUTCOMES:
Change from baseline of central spinal fluid heparan sulfate after treatment | 24 months
Change from baseline of plasma or urine glycosaminoglycans or heparan sulfate after treatment | 24 Months
Change from baseline in CSF or plasma NAGLU enzyme activity levels after treatment | 24 Months
Change from baseline in liver and/or spleen volumes after treatment, as measured by magnetic resonance imaging | 24 Months
Change from baseline in brain volumes after treatment, as measured by magnetic resonance imaging | 24 Months
Change from baseline in the Cognitive Age Equivalent (Developmental Age) compared to Natural History Study, calculated using the Bayley Scales of Infant and Toddler Development or the Kaufman Assessment Battery for Children | 24 Months
Change from baseline in the Adaptive Age Equivalent score after treatment compared to Natural History Study data, as assessed by parent report using the Vineland Adaptive Behavior Scale II Survey form | 24 Months
Change from baseline Developmental Quotient after treatment compared to Natural History Study data assessed by the Mullen Scales of Early Learning or the Kaufman Assessment Battery for Children. | 24 Months
Change from baseline in Pediatric Quality of Life Inventory (PedsQL™) Generic Core Scales total score | 24 Months
Change from baseline in parent quality of life, using the Parenting Stress Index, 4th Edition (PSI-4) short form | 24 Months
Determination of vector shedding analysis in plasma, saliva, urine and feces will provide preliminary data for the Environmental Risk Assessment | 24 Months

CONTACTS AND LOCATIONS:
Locations (4):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- Armand-Trousseau Hospital, Paris, France
- University Hospital Hamburg-Eppendorf, Hamburg, Germany
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data

REFERENCES:
- [Background] Fu H, Dirosario J, Killedar S, Zaraspe K, McCarty DM. Correction of neurological disease of mucopolysaccharidosis IIIB in adult mice by rAAV9 trans-blood-brain barrier gene delivery. Mol Ther. 2011 Jun;19(6):1025-33. doi: 10.1038/mt.2011.34. Epub 2011 Mar 8. PMID 21386820
- [Background] Truxal KV, Fu H, McCarty DM, McNally KA, Kunkler KL, Zumberge NA, Martin L, Aylward SC, Alfano LN, Berry KM, Lowes LP, Corridore M, McKee C, McBride KL, Flanigan KM. A prospective one-year natural history study of mucopolysaccharidosis types IIIA and IIIB: Implications for clinical trial design. Mol Genet Metab. 2016 Nov;119(3):239-248. doi: 10.1016/j.ymgme.2016.08.002. Epub 2016 Aug 18. PMID 27590925
- [Background] Neufeld EF, Cantz MJ. Corrective factors for inborn errors of mucopolysaccharide metabolism. Ann N Y Acad Sci. 1971 Jul 6;179:580-7. doi: 10.1111/j.1749-6632.1971.tb46934.x. No abstract available. PMID 4255108
- [Background] Weber B, Guo XH, Kleijer WJ, van de Kamp JJ, Poorthuis BJ, Hopwood JJ. Sanfilippo type B syndrome (mucopolysaccharidosis III B): allelic heterogeneity corresponds to the wide spectrum of clinical phenotypes. Eur J Hum Genet. 1999 Jan;7(1):34-44. doi: 10.1038/sj.ejhg.5200242. PMID 10094189
- [Background] Wijburg FA, Wegrzyn G, Burton BK, Tylki-Szymanska A. Mucopolysaccharidosis type III (Sanfilippo syndrome) and misdiagnosis of idiopathic developmental delay, attention deficit/hyperactivity disorder or autism spectrum disorder. Acta Paediatr. 2013 May;102(5):462-70. doi: 10.1111/apa.12169. Epub 2013 Feb 6. PMID 23336697
- [Background] de Ruijter J, Valstar MJ, Wijburg FA. Mucopolysaccharidosis type III (Sanfilippo Syndrome): emerging treatment strategies. Curr Pharm Biotechnol. 2011 Jun;12(6):923-30. doi: 10.2174/138920111795542651. PMID 21235449
- [Background] Murrey DA, Naughton BJ, Duncan FJ, Meadows AS, Ware TA, Campbell KJ, Bremer WG, Walker CM, Goodchild L, Bolon B, La Perle K, Flanigan KM, McBride KL, McCarty DM, Fu H. Feasibility and safety of systemic rAAV9-hNAGLU delivery for treating mucopolysaccharidosis IIIB: toxicology, biodistribution, and immunological assessments in primates. Hum Gene Ther Clin Dev. 2014 Jun;25(2):72-84. doi: 10.1089/humc.2013.208. Epub 2014 Apr 10. PMID 24720466
- [Background] Ribera A, Haurigot V, Garcia M, Marco S, Motas S, Villacampa P, Maggioni L, Leon X, Molas M, Sanchez V, Munoz S, Leborgne C, Moll X, Pumarola M, Mingozzi F, Ruberte J, Anor S, Bosch F. Biochemical, histological and functional correction of mucopolysaccharidosis type IIIB by intra-cerebrospinal fluid gene therapy. Hum Mol Genet. 2015 Apr 1;24(7):2078-95. doi: 10.1093/hmg/ddu727. Epub 2014 Dec 18. PMID 25524704
- [Background] Hamano K, Hayashi M, Shioda K, Fukatsu R, Mizutani S. Mechanisms of neurodegeneration in mucopolysaccharidoses II and IIIB: analysis of human brain tissue. Acta Neuropathol. 2008 May;115(5):547-59. doi: 10.1007/s00401-007-0325-3. Epub 2007 Dec 4. PMID 18060551
- [Background] Tamagawa K, Morimatsu Y, Fujisawa K, Hara A, Taketomi T. Neuropathological study and chemico-pathological correlation in sibling cases of Sanfilippo syndrome type B. Brain Dev. 1985;7(6):599-609. doi: 10.1016/s0387-7604(85)80008-5. PMID 3938624
- [Background] Mingozzi F, High KA. Immune responses to AAV in clinical trials. Curr Gene Ther. 2011 Aug;11(4):321-30. doi: 10.2174/156652311796150354. PMID 21557723
- [Background] Saeki I, Tokunaga S, Matsuura T, Hayashida M, Yanagi Y, Taguchi T. A formula for determining the standard liver volume in children: a special reference for neonates and infants. Pediatr Transplant. 2012 May;16(3):244-9. doi: 10.1111/j.1399-3046.2011.01624.x. Epub 2011 Dec 12. PMID 22151603
- [Background] Schlesinger AE, Edgar KA, Boxer LA. Volume of the spleen in children as measured on CT scans: normal standards as a function of body weight. AJR Am J Roentgenol. 1993 May;160(5):1107-9. doi: 10.2214/ajr.160.5.8470587.
- [Background] Malm G, Mansson JE. Mucopolysaccharidosis type III (Sanfilippo disease) in Sweden: clinical presentation of 22 children diagnosed during a 30-year period. Acta Paediatr. 2010 Aug;99(8):1253-7. doi: 10.1111/j.1651-2227.2010.01800.x. Epub 2010 Mar 14. PMID 20337777
- [Background] Dale DC, Fauci AS, Guerry D IV, Wolff SM. Comparison of agents producing a neutrophilic leukocytosis in man. Hydrocortisone, prednisone, endotoxin, and etiocholanolone. J Clin Invest. 1975 Oct;56(4):808-13. doi: 10.1172/JCI108159. PMID 1159089
- [Background] Summers C, Rankin SM, Condliffe AM, Singh N, Peters AM, Chilvers ER. Neutrophil kinetics in health and disease. Trends Immunol. 2010 Aug;31(8):318-24. doi: 10.1016/j.it.2010.05.006. PMID 20620114
- [Derived] McCurdy VJ, Johnson AK, Gray-Edwards HL, Randle AN, Bradbury AM, Morrison NE, Hwang M, Baker HJ, Cox NR, Sena-Esteves M, Martin DR. Therapeutic benefit after intracranial gene therapy delivered during the symptomatic stage in a feline model of Sandhoff disease. Gene Ther. 2021 Apr;28(3-4):142-154. doi: 10.1038/s41434-020-00190-1. Epub 2020 Sep 3. PMID 32884151